CLINICAL TRIAL: NCT07141693
Title: Renal Oximetry-Guided Anesthesia With Near-Infrared Spectroscopy for Improved Postoperative Outcomes in Hepatectomy: A Dual-Center, Prospective, Randomized, Single-Blind Investigator-Initiated Pilot Trial
Brief Title: Renal Oximetry-Guided Anesthesia With Near-Infrared Spectroscopy for Improved Postoperative Outcomes
Acronym: ROGAR
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Beijing Tsinghua Changgeng Hospital (Other)
Responsible Party: Principal Investigator, Hao Li, Prof, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ChinesePLA_ROGAR_Pilot
Record Dates: First submitted 2025-08-09; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- NIRS-guided anesthesia management group (Experimental): NIRS-guided management where a predefined 6-step intervention protocol (volume optimization, vasoactive drugs, inotropes, heart rate management, transfusion, and FiO₂ increase)
  Interventions: Procedure: NIRS-guided management
- Standard anesthesia management (Placebo Comparator): standard anesthesia management
  Interventions: Procedure: Standard anesthesia management

INTERVENTIONS:
Procedure: NIRS-guided management — NIRS-guided management where a predefined 6-step intervention protocol (volume optimization, vasoactive drugs, inotropes, heart rate management, transfusion, and FiO₂ increase)
  Arms: NIRS-guided anesthesia management group
Procedure: Standard anesthesia management — Standard anesthesia management
  Arms: Standard anesthesia management

SUMMARY:
The trial is a prospective, randomized, single-blind, pilot study investigating whether near-infrared spectroscopy (NIRS)-guided optimization of intraoperative renal oxygen saturation (SrtO₂) reduces postoperative acute kidney injury (AKI) in patients undergoing elective hepatectomy. The trial will enroll 80 adults (≥45 years, American society of Aneshesiologists physical status I-III), randomizing them to either standard anesthesia management or NIRS-guided management where a predefined 6-step intervention protocol (volume optimization, vasoactive drugs, inotropes, heart rate management, transfusion, and FiO₂ management) is triggered if SrtO₂ decreases >10% from baseline. Primary outcomes are the incidence of AKI within 7 days and the 28-day Comprehensive Complication Index (CCI). The study aims to determine if real-time SrtO₂ monitoring and proactive intervention can prevent this serious complication, based on previous observational data linking renal desaturation to AKI risk.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 45 years
* Scheduled for elective hepatectomy
* Planned for general anesthesia with endotracheal intubation
* BMI < 30 kg/m2
* Preoperative ultrasound shows renal cortical to skin distance ≤ 4 cm
* ASA classification I-III
* Consenting to participate and signing informed consent

Exclusion Criteria:

* Liver transplantation surgery
* Preoperative renal dysfunction or requirement for dialysis treatment;
* Contraindications to vasoactive drugs such as norepinephrine or dopamine as determined by the clinician;
* Severe cardiopulmonary insufficiency (severe arrhythmia, heart failure, respiratory failure, chronic obstructive pulmonary disease), or a serious cardiovascular or cerebrovascular event within the last six months before randomization (such as acute heart failure, acute myocardial infarction, stroke, etc.);
* Patient refusal to participate or current participation in another experimental study;
* Other factors deemed unsuitable for inclusion by the researcher.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Actue kidney injury | Postoperative Day 1-7
  An increase in serum creatinine of ≥26.5 μmol/L from baseline within 48 hours or an increase of ≥50% from baseline within 7 days
Comprehensive Complication Index | Postoperative Day 1-28
  The co-primary outcome is the Comprehensive Complication Index (CCI) score, which includes all complications occurring from randomization to the 28-day follow-up period and calculated using the Clavien-Dindo classification (CDC).

SECONDARY OUTCOMES:
Total duration and proportion of time during surgery of renal desaturation | Intraoperative
  Total duration and proportion of time during surgery when renal oxygen saturation decreases by >10% from baseline
Area under the curve for renal oxygen desaturation | Intraoperative
  Area under the curve for renal oxygen saturation decrease by >10% from baseline
Use of vasoactive drugs | Intraoperative
  The type and total dose of vasoactive drugs
Intraoperative blood pressure levels | Intraoperative
  Intraoperative low blood pressure and the lowest level
AKI grading | Postoperative Day 1-7
  According to serum creatinine level to conduct AKI grade
Overall incidence of postoperative complications | Postoperative Day 1-28
  Overall incidence of postoperative complications, including neurological, respiratory, cardiovascular complications, acute kidney injury, and sepsis.
mortality | Postoperative Day 1-28
  In-hospital mortality and 28-day postoperative mortality

IPD SHARING:
Plan to Share IPD: No